CLINICAL TRIAL: NCT06469359
Title: Development of a Methodology to Analyze Nasal Tissue-resident Memory Immune Cells and Peripheral Memory Cells Able to Migrate to Airway Tissues (MUCOVAC)
Brief Title: Analyzes of Nasal Tissue-resident Memory Immune Cells and Peripheral Memory Cells Able to Migrate to Airway Tissues (MUCOVAC)
Acronym: MUCOVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 23CH294; 2024-A00255-42 (Other: ANSM)
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
Keywords: Nasal immune cells; sampling device; airway immunity; memory immune responses; T cells; B cells
MeSH Terms: interventions — Blood Specimen Collection; Neutralization Tests; Enzyme-Linked Immunospot Assay

STUDY DESIGN:
Intervention Model Description: Prospective study in healthy volunteers. Randomized, single-blind, cross-over trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FLOQSwab, Copan Diagnostics (Experimental): Nasal cells are collected in both nostrils using one FLOQSwab per nostril
  Interventions: Device: Nasal tissue-resident memory T and B cells; Device: Nasal fluid sampling; Device: Saliva sampling; Other: Blood sampling; Diagnostic Test: ELISA; Diagnostic Test: Neutralization test; Diagnostic Test: ELISPot; Diagnostic Test: Transcriptomics
- Rhino-Pro Curette, Arlington Scientific (Experimental): Nasal cells are collected in both nostrils using one curette per nostril
  Interventions: Device: Nasal tissue-resident memory T and B cells; Device: Nasal fluid sampling; Device: Saliva sampling; Other: Blood sampling; Diagnostic Test: ELISA; Diagnostic Test: Neutralization test; Diagnostic Test: ELISPot; Diagnostic Test: Transcriptomics
- Cervical brush, Microm Microtech (Experimental): Nasal cells are collected in both nostrils using one brush per nostril
  Interventions: Device: Nasal tissue-resident memory T and B cells; Device: Nasal fluid sampling; Device: Saliva sampling; Other: Blood sampling; Diagnostic Test: ELISA; Diagnostic Test: Neutralization test; Diagnostic Test: ELISPot; Diagnostic Test: Transcriptomics

INTERVENTIONS:
Device: Nasal tissue-resident memory T and B cells — Nasal tissue-resident memory T and B cells are quantified using flow cytometry.
Device: Nasal fluid sampling — Nasal fluid is collected using strip (Hunt Development) in both nostrils
Device: Saliva sampling — Saliva is collected using Oracol (Malvern Medical Developments)
Other: Blood sampling — Isolation of peripheral blood mononuclear cells (PBMC) and serum from blood
Diagnostic Test: ELISA — ELISA to measure antibody responses in mucosal fluids and blood
Diagnostic Test: Neutralization test — Neutralization test to measure neutralizing antibody responses in mucosal fluids and blood to measure neutralizing antibody responses in mucosal fluids and blood
Diagnostic Test: ELISPot — ELISPot to measure cellular responses in blood
Diagnostic Test: Transcriptomics — Transcriptomics to quantify the gene expression of immunological markers in blood

SUMMARY:
Clinical evaluation of vaccines against respiratory viruses is currently based on the analysis of systemic immune responses, whereas respiratory immunity is the first line of defense against respiratory pathogens. In addition to secretory immunoglobulin A (IgA) in mucosal fluids which are essential to neutralize the pathogens at mucosal surfaces, tissue-resident memory immune cells have been shown to be crucial in protection. Furthermore, memory immune cells in blood able to migrate to airway tissues also play a crucial role. Airway immune responses have not been studied a lot due to the lack of a standardized methodology to evaluate them in humans.

DETAILED DESCRIPTION:
The goal of this study is to develop a methodology to collect and analyze nasal tissue-resident memory T and B cells and to evaluate peripheral memory T and B cells expressing airway homing markers in healthy volunteers. Three devices for nasal cell sampling will be compared. Tissue-resident and peripheral memory immune responses will be determined using flow cytometry and correlated with humoral and cellular responses, as well as with gene expression at mucosal and systemic levels. .

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to the Social Security System
* Signed informed consent form

Exclusion Criteria:

* History of recurrent nosebleeds or systemic hemorrhages
* Previous injury or surgery which modified nasal cavity (e.g. deviated nasal septum)
* Individuals receiving anticoagulant therapy
* Individuals who experienced a severe respiratory infection leading to hospitalization in the last 6 months
* Individuals who received an antibiotic therapy for respiratory infection or any other infection in the last 6 months
* Immunocompromised individuals, or individuals taking immunosuppressed therapy or having a pathology (chronic infection, auto-immune disease) which could impact on immunity based on investigator's opinion
* Unstable chronic pathology
* People deprived of liberty or hospitalized without any consent
* People under guardianship (authorship or curators)
* Individuals who received a vaccine (any vaccine) in the last 30 days
* Pregnant or breast-feeding people
* Individuals experiencing respiratory infection symptoms. Inclusion will be postponed up to 7 days after the symptom resolution

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Frequency of resident memory lymphocytes in the nasal mucosa measured by FLOQSwab | At inclusion, one month, two months
  This outcome is measured by the three devices :
  * FLOQSwab
  * Rhino-Pro Curette
  * Cervical brush

SECONDARY OUTCOMES:
Frequencies of resident memory T and B lymphocytes | At inclusion, one month, two months
  Frequencies of resident memory T and B lymphocytes are measured by the three devices :
  * FLOQSwab
  * Rhino-Pro Curette
  * Cervical brush
Expression levels of respiratory mucosal migration markers on peripheral memory lymphocytes | At inclusion, one month, two months
  This outcome is measured by the three devices :
  * FLOQSwab
  * Rhino-Pro Curette
  * Cervical brush
Visual analog scale for pain | At inclusion, one month, two months
  Scale from 0 to 10 (0 = no pain, 10 = intolerable pain)
  This outcome is measured by the three devices :
  * FLOQSwab
  * Rhino-Pro Curette
  * Cervical brush

CONTACTS AND LOCATIONS:
Overall Officials: ELISABETH BOTELHO-NEVERS, MD-PhD, Principal Investigator — CHU DE SAINT-ETIENNE; STEPHANE PAUL, MD-PhD, Study Director — CHU de Saint-Etienne; STEPHANIE LONGUET, PhD, Study Chair — Université de Saint-Etienne
Locations (1):
- Centre Hospitalier Universitaire, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No